CLINICAL TRIAL: NCT05045547
Title: Expanding the Roles of Village Malaria Workers: Operational Research in Cambodia
Brief Title: Village Malaria Worker Expansion
Acronym: CAM-VMW
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: HCR21005
Record Dates: First submitted 2021-06-01; First posted 2021-09-16 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Febrile Illness
Keywords: Febrile Illness; Village Health Worker; Cambodia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with febrile illness: Febrile patients attending village malaria workers (VMWs)
- Health centre staffs: Health centre staffs from 12 rural health centres
- Key stakeholders: Key stakeholders , for example health managers and health professionals:
  * the director, deputy-directors, and technical officers at the National Malaria Control Program;
  * the directors and deputy-directors of the Provincial Health Departments in Battambang and Pailin province;
  * health officers actively involved in community-based (malaria) programmes at the district levels in Battambang and Pailin provinces;
  * health workers (i.e., nurses or doctors) actively involved in community-based (malaria) programmes in Battambang and Pailin provinces;
  * community representatives and village malaria workers from villages in both Battambang Pailin province.

SUMMARY:
This project will conduct pragmatic operational research in rural communities served by approximately 12 health centres and 120 village malaria workers in Battambang/Pailin, western Cambodia.

This study is funded by Global Fund/Regional Artemisinin Initiative (RAI3E). The grant reference number is QSE-M-UNOPS-MORU-20864-007-42

DETAILED DESCRIPTION:
This is an integration of activities with the South and Southeast Asian Community-based Trials Network (SEACTN) that is ongoing in Lao PDR and Bangladesh. The SEACTN study aims to identify the most relevant ways in which village health worker roles can be expanded to include management of community febrile illness. A number of SEACTN activities will also be conducted in Cambodia alongside this project.

For this project, the study team will test specific examples of expanded roles of VMWs including testing for other causes of fever in people who are malaria negative and assessing the feasibility of diagnostics other than malaria RDTs at health centres. Quantitative and qualitative data will be collected to determine acceptability, a mixed-methods approach will be used for the assessment:

• Quantitative method

Participants with febrile illness attending village malaria workers will be tested by novel rapid diagnostic tests (Dengue and CRP rapid test) in addition to a standard malaria test. Village malaria workers (VMWs)/ mobile malaria workers (MMWs) will be trained to conduct a package of activities ((i) hygiene and sanitation; (ii) disease surveillance; (iii) EPI and ANC support; (iv) management of mild common illnesses that they will carry out alongside their usual role of testing (RDTs) and treating malaria. If possible, within a week of conducting a novel RDT, a well-being follow up will be undertaken by the VMW, either via telephone or face-to-face. For the primary outcomes, the study team will report numbers and proportions of training modules passed, malaria tests performed, new diagnostic tests performed correctly, algorithms followed correctly, number of consultations, coverage estimates, and the study team will use the national malaria information system to provide a comparison in activity levels compared to other areas of Cambodia. The study team will record the incidence and aetiology of febrile illnesses.

• Qualitative method

A set of interviews/discussions with health centre staffs and local stakeholders will be conducted to refine the intervention design and implementation strategy. To this end, the interviews will elicit the views and experience of local stakeholders on (1) health care needs and gaps in local communities, (2) views and past experiences concerning the implementation of the VMW programme, with a focus on challenges and good practices around the use of RDTs, and (3) their views about suitable methods and strategies to expand the current VMW programme considering the new technologies available.

Findings from the study will highlight to the wider scientific community the benefits and challenges of expanding the roles of VMW/MMWs.

ELIGIBILITY:
Inclusion Criteria

1. Quantitative research

   * Written informed consent
   * Willingness to provide blood sample
   * Fever (≥37.5 C) or history of fever within 24 hours
2. Qualitative research

2.1 Health centre-based evaluation of novel diagnostics

* Health centre staff who have received training in the use of the novel diagnostics used in the study
* Willing and able to give informed consent for participation in the study

2.2 Stakeholder analysis

* Adults, male or female, aged 18 years and over
* Willing and able to give informed consent for participation in the study

Exclusion Criteria

1. Quantitative research

   • Participants requires urgent medical attention
2. Qualitative research

   * Identified with intellectual and/or cognitive disability
   * History of or current psychiatric illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Quantitative research
     Participants: Febrile patients attending village malaria workers (VMWs)
  2. Qualitative research
  2.1 Health centre-based evaluation of novel diagnostics
  Participants: Health centre staffs from 12 rural health centres
  2.2 Stakeholder analysis
  Participants: Key stakeholders , for example health managers and health professionals:
  * the director, deputy-directors, and technical officers at the National Malaria Control Program;
  * the directors and deputy-directors of the Provincial Health Departments in Battambang and Pailin province;
  * health officers actively involved in community-based (malaria) programmes at the district levels in Battambang and Pailin provinces;
  * health workers (i.e., nurses or doctors) actively involved in community-based (malaria) programmes in Battambang and Pailin provinces;
  * community representatives and village malaria workers from villages in both Battambang Pailin province.
Sampling Method: Non-Probability Sample
Enrollment: 7191 (Actual)
Dates: Start 2022-04-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The number of VMW consultations by patients | Approximately 18-24 months
  The number of VMW consultations by patients with a febrile and/or non-febrile illness along with the number of malaria RDTs used will be recorded. Comparing these data across the different intervention packages introduced for VMWs.

SECONDARY OUTCOMES:
The number of VMWs that can correctly perform RDTS following a directly observed practical assessment and questionnaire. | Approximately 18-24 months
  The number of VMWs that can correctly perform RDTS following a directly observed practical assessment and questionnaire.
The number of VMWs who correctly follow the treatment algorithms following a directly observed practical assessment and questionnaire. | Approximately 18-24 months
  The number of VMWs who correctly follow the treatment algorithms following a directly observed practical assessment and questionnaire.
The overall consensus of stakeholders regarding the new roles of VMWs following stakeholder interviews | 0 months, mid-point of the study (12 months) and at study completion (24 months)
  The overall consensus of stakeholders regarding the new roles of VMWs following stakeholder interviews
The overall consensus of stakeholders of the impact on non-malarial febrile illness management following stakeholder interviews | 0 months, mid-point of the study (12 months) and at study completion (24 months)
  The overall consensus of stakeholders of the impact on non-malarial febrile illness management following stakeholder interviews
The number of VMWs that can correctly deliver one of four health intervention packages following a directly observed practical assessment and questionnaire. | 0 months, mid-point of the study (12 months) and at study completion (24 months)
  The number of VMWs that can correctly deliver one of four health intervention packages following a directly observed practical assessment and questionnaire.
The number of health centre staff that can correctly perform RDTs following a directly observed practical assessment and questionnaire | Approximately 18-24 months
  The number of health centre staff that can correctly perform RDTs following a directly observed practical assessment and questionnaire
The overall consensus of stakeholders on the use of novel RDTs following stakeholder interviews and focus group discussions. | Approximately 18-24 months
  The overall consensus of stakeholders on the use of novel RDTs following stakeholder interviews and focus group discussions.
The overall consensus of stakeholders regarding these new roles following stakeholder interviews | At study completion (24 months)
  The overall consensus of stakeholders regarding these new roles following stakeholder interviews

OTHER OUTCOMES:
The number of patients appropriately referred for further care | Approximately 18-24 months
  The number of patients appropriately referred for further care

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Peto, Dr., Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit; James J Callery, Dr., Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Action for Health and Development, Battambang, Cambodia

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be under the custodianship of MORU. With participant's consent, data from this study may be shared in a de-identified form with other groups or researchers in accordance with the MORU Data Sharing Policy.
Time Frame: After completion of trial activities and reporting
Access Criteria: MORU Data Sharing Policy. (http://www.tropmedres.ac/data-sharing-policy)